CLINICAL TRIAL: NCT06966609
Title: Additional Effects of Cuevas Medek Exercises Along With Conventional Physical Therapy on Gross Motor Proficiency and Quality of Life, in Children With Spastic Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/36
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Spastic Diplegia Cerebral Palsy; Quality of Lifte; Motor Function
Keywords: Spastic Diplegic Cerebral Palsy; Gross motor proficiency; quality of life
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group A (Experimental): It includes participants receiving cuevas medek exercise combined with conventional physical therapy for 12 weeks treatment.
  1. Stretching Exercises (PNF stretching)
     * 0-6 weeks; 3 sets (5 repetition of 20sec) 4 times a week
     * 6-12 weeks; 3 sets(10 repetition of 60sec) 4 times a week
     * Muscles included:
     Flexors (hip, knee, ankle), extensors (hip, knee, ankle), abductor(hip) and adductors(hip)
  2. Strengthening Exercises (Isometric muscle strengthening )
     * 3 sets ( 10 repetition)
     * Rest interval: 1min
     * Frequency: 3 times a week
     * Muscles included:
  Flexors(hip, knee, ankle), extensors(hip, knee, ankle), abductor(hip) and adductors(hip) 3. Gait training Parallel bar walking 4. Cuevas Medek Exercise(99 exercises)
  * Frequency: 3 times a week
  * Duration: 45mins
  * Repetition: 3-8 times
  * Exercises divided into following, will be administered according to patient need/goal;
    1. Head control
    2. Trunk control
    3. Trunk and hip control
    4. Coordination
    5. Balance reaction
    6. Stability
  Interventions: Procedure: Experimental Group
- Interventional Group B (Active Comparator): It includes participants receiving conventional physical therapy for 12 weeks treatment.
  1. Stretching Exercises (PNF stretching)
     * 0-6 weeks; 3 sets (5 repetition of 20sec) 4 times a week
     * 6-12 weeks; 3 sets(10 repetition of 60sec) 4 times a week
     * Muscles included:
     Flexors (hip, knee, ankle), extensors (hip, knee, ankle), abductor(hip) and adductors(hip)
  2. Strengthening Exercises (Isometric muscle strengthening )
     * 3 sets ( 10 repetition)
     * Rest interval: 1min
     * Frequency: 3 times a week
     * Muscles included:
     Flexors(hip, knee, ankle), extensors(hip, knee, ankle), abductor(hip) and adductors(hip)
  3. Gait training Parallel bar walking Treatment time: 45mins
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Control Group — Conventional Physical Therapy ( 12 weeks intervention) 24 randomly allocated participants will get the conventional physical therapy that includes the stretching exercises (PNF technique) for 6 weeks; targeting all the affected lower limb muscles, strengthening exercises of all the weak lower limb muscles for 12 weeks along with gait training on parallel bars. Duration of session is 45 min.
  Arms: Interventional Group B
Procedure: Experimental Group — Conventional Physical Therapy and Cuevas Medek Exercises ( 12 weeks intervention) 24 randomly allocated participants will get the conventional physical therapy that includes the stretching exercises (PNF technique) for 6 weeks; targeting all the affected lower limb muscles, strengthening exercises of all the weak lower limb muscles for 12 weeks along with gait training on parallel bars.Along with conventional physical therapy, experimental group participants will get Cuevas Medek Exercises that includes antigravity exercises, specefic types of stretchings and balancing exercises. Types of exercises that will be performed on the patient out of 100 exercises,will depend on the patient's need that is affecting his or her gross motor proficiency.Total duration of session is 90 min.
  Arms: Interventional Group A

SUMMARY:
Cerebral palsy (CP) is a prevalent pediatric neurological disorder hindering movement and posture development due to non-progressive disruptions in brain development. Motor disorders along with dysfunctions in sensations, perception, cognition, communication, behavior and secondary musculoskeletal problems are also present in children with CP.

Cuevas Medek Exercises (CME) is an innovative, intensive and dynamic therapy approach for management of movement disorders. It evoke automatic postural responses in children with motor delay problems by application of distal support, triggering stronger gravity induced reactions to enhanced motor output by compelling both mind and body responses.

It incorporates antigravity posture, ROM, weight-bearing, and stretching into functional exercises; for improved agility, flexibility, balance and coordination.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the additional effect of Cuevas Medek Exercises with conventional exercises on gross motor proficiency in children with spastic diplegic cerebral palsy.
2. To determine the additional effect of Cuevas Medek Exercises with conventional exercises on quality of life of caregiver and children with spastic diplegic cerebral palsy.

HYPOTHESIS:

Alternate Hypothesis:

1. There is a statistically significant effect of Cuevas Medek Exercises in conjunction with conventional physical therapy as compared to conventional physical therapy alone on gross motor proficiency in children with spastic diplegic cerebral palsy. (p<0.05)
2. There is a statistically significant effect of Cuevas Medek Exercises in conjunction with conventional physical therapy as compared to conventional physical therapy alone on quality of life in children with spastic diplegic cerebral palsy. (p<0.05)

Null Hypothesis:

1. There is a statistically no significant effect of Cuevas Medek Exercises in conjunction with conventional physical therapy as compared to conventional physical therapy alone on gross motor proficiency in children with spastic diplegic cerebral palsy. (p>0.05)
2. There is a statistically no significant effect of Cuevas Medek Exercises in conjunction with conventional physical therapy as compared to conventional physical therapy alone on quality of life in children with spastic diplegic cerebral palsy. (p>0.05)

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Fauji Foundation Hospital Study duration 1 year following synopsis approval.(Feb 2024- Jan 2025)

Selection Criteria:

Inclusion Criteria

* diagnosed spastic diplegic cerebral palsy children
* age group 6-12 years old
* both male and female
* GMFCS II & III
* parents of spastic diplegic CP child

Exclusion Criteria

* diagnosed cognitive impairment
* diagnosed hearing impairment and visual impairment
* children with planned surgical procedures during study period

Sampling technique: convenicence sampling

Outcome Measures:

1. Gross motor function measure
2. CP QOL - CHILD

Data analysis techniques:

Data will be analyzed using SPSS version 20.0.0.

Significance of the study:

* Till date no study has yet evaluated the effect of Cuevas Medek Exrcises on gross motor proficiency and quality of life in children with spastic diplegic cerebral palsy. Therefore, advancement in the scientific knowledge can be achieved.
* Caregivers of cerebral palsy suffer from a substantial psychosocial burden. Therefore, to determine whether CME Therapy effects functional dependency and quality of life of both patient and caregivers.
* This study will contribute to future research directions and encouraging further exploration of CME Therapy as a promising intervention for spastic diplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed spastic diplegic cerebral palsy children
* age group 6-12 years old
* both male and female
* GMFCS II & III
* parents of spastic diplegic CP child

Exclusion criteria:

* diagnosed cognitive impairment
* diagnosed hearing impairment and visual impairment
* children with planned surgical procedures during study period

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function | 12 weeks
  Gross Motor Function Measure-88 score, will be used to assess gross motor function in children with cerebral palsy. It is a four point scale, consists of 88 items divided into five dimensions of gross motor function: a. lying and rolling, b. crawling and kneeling, c. sitting, d. standing, e. walking, running and jumping. It takes about 45 to 60 minutes. Equipments required for this measure tool are; mat, bench, toy and access to stairs.
  Item scores are summed to calculate raw and percent scores for each of the five dimensions. Then, Average the percent scores for each dimension to get the total score. Total score (in percent), will be compared on each assessment to find out the improvement in the individual through that specefic intervention.
Quality of Life | 12 weeks
  CP QOL Child Primary Caregiver It is a validated questionnaire that assesses the subjective well- being and happiness of children with CP. It consist of 66 questions and should be answered by caregivers of CP child, who report their perception of their child's quality of life of areas: well being and social acceptance, functionality, participation and physical health, emotional well being and self esteem, access to services, pain and disability impact and family health. The questionnaire is scored by summing the items to get a total score, with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan